CLINICAL TRIAL: NCT02788747
Title: A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effects of Multiple Subcutaneous Injections of Elamipretide on Left Ventricular Function in Subjects With Stable Heart Failure With Reduced Ejection Fraction
Brief Title: Effect of Elamipretide on Left Ventricular Function in Subjects With Stable Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPIHF-201; 2014-005724-10 (EudraCT Number)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 mg elamipretide (Experimental): 4 mg elamipretide once daily for 28 consecutive days
  Interventions: Drug: 4 mg elamipretide
- 40 mg elamipretide (Experimental): 40 mg elamipretide once daily for 28 consecutive days
  Interventions: Drug: 40 mg elamipretide
- Placebo (Placebo Comparator): Placebo once daily for 28 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4 mg elamipretide — Subcutaneous injection of 4 mg elamipretide administered once daily for 28 consecutive days
  Other Names: MTP-131; Bendavia
  Arms: 4 mg elamipretide
Drug: 40 mg elamipretide — Subcutaneous injection of 40 mg elamipretide administered once daily for 28 consecutive days
  Other Names: MTP-131; Bendavia
  Arms: 40 mg elamipretide
Drug: Placebo — Subcutaneous injection of placebo administered once daily for 28 consecutive days
  Arms: Placebo

SUMMARY:
This was a randomized, double-blinded, placebo-controlled, multiple-dose study in subjects with stable heart failure (HF) with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
This was a randomized, double-blinded, placebo-controlled, multiple-dose study in subjects with stable heart failure (HF) with reduced ejection fraction (HFrEF). After completing the Screening period, a total of 71 subjects were randomized, in a 1:1:1 ratio, to receive either placebo, 4 mg elamipretide, or 40 mg elamipretide once daily for 28 consecutive days.

Each treatment group went through 3 distinct periods: Screening, Treatment, and Follow up.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent form (ICF) prior to participation in any study-related procedures.
* Age ≥40 and ≤80 years.
* A known history of chronic ischemic or non-ischemic cardiomyopathy of at least 6 months duration from the time of the initial diagnosis.
* Receiving heart failure (HF) treatment, including, but not limited to, angiotensin converting enzyme inhibitors (ACEI) and/or angiotensin receptor blockers (ARB), and an evidence-based beta blocker for the treatment of HF. Subjects who cannot tolerate ACEI or ARB due to reduced renal function or hypotension are eligible. Subjects may be receiving aldosterone antagonists, but this is not a requirement for the study.
* HF is considered to be stable in the judgment of the Investigator AND doses of HF treatment have been stable for at least 1 month prior to the Screening Visit.
* In normal sinus rhythm (electrocardiogram documented) at Screening and Day 1 and no history of atrial fibrillation in the past 12 months
* No hospitalization related to HF within 1 month prior to the Screening Visit.
* Left Ventricular Ejection Fraction (LVEF) ≤ 40% by 2-D echocardiography at Screening.
* At least 3 viable segments (hyperenhancement ≤ 25%) by a qualifying delayed gadolinium-enhanced cardiac MRI examination at Screening (confirmed by independent core lab).
* Women of childbearing potential must agree to use 1 of the following methods of birth control from the date they sign the ICF until two months after the last dose of study medication:

  * Abstinence, maintenance of monogamous relationship with a male partner who has been surgically sterilized by vasectomy, or barrier method AND either hormonal contraception or an intrauterine device or system.

Exclusion Criteria:

* History of any concurrent medical condition which, in the opinion of the Investigator, significantly increased the potential risks associated with administration of study medication or any other aspect of study participation.
* Any contraindication to MRI scanning.
* Left ventricular end diastolic dimension (LVEDD) indexed to Body Surface Area is > 45 mm/m2.
* Coronary or peripheral revascularization procedures, valvular procedures, OR any major surgical procedure within 3 months prior to the Screening Visit.
* Acute coronary syndrome, stroke or transient ischemic attack (TIA) within 3 months prior to the Screening Visit.
* Obstructive or restrictive cardiomyopathy, infiltrative diseases of the myocardium (e.g., amyloid, sarcoid, etc.) myocarditis, or reductions in LV function thought to be secondary primarily to valvular heart disease, prior cardiac valve surgery or known aortic stenosis.
* The presence or anticipated placement of any pacemaker, implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy (CRT) devices during the ensuing 6-week study period.
* Presence of second degree or advanced heart block.
* Uncontrolled hypertension defined as a systolic blood pressure > 160 mmHg or a diastolic blood pressure > 110 mmHg on at least two consecutive readings.
* Presence of any left ventricular thrombus, pericardial disease, uncorrected thyroid disease or a dyskinetic left ventricular aneurysm.
* History of cancer that causes symptoms, disabilities, or is likely to lead to hospitalization or treatment in the next 12 months.
* Currently receiving treatment with chemotherapeutic agents or immunosuppressant agents or has received prior radiation therapy to the chest.
* Liver enzymes (alanine aminotransferase [ALT] AND/OR aspartate. aminotransferase [AST]) elevation > 3 times the upper limit of normal (ULN).
* Total bilirubin > 1.5 times ULN in the absence of Gilbert's Syndrome.
* Bleeding diathesis or any known blood dyscrasia.
* Anemia, defined as hemoglobin < 9 g/dL or planned blood transfusions in the next 6 weeks.
* Estimated glomerular filtration rate (eGFR) < 30 mL/min, using the Modification of Diet in Renal Disease (MDRD) Study equation.
* History of hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) infection, or diagnosis of immunodeficiency.
* Known active drug or alcohol abuse within 1 year of the Screening Visit. Alcohol abuse is defined as 15 or more drinks for men per week or 8 or more for women.
* Recipient of any investigational drugs, stem cell or gene therapies, or devices OR participation in another clinical trial, within 3 months prior to the Screening Visit.
* Female subjects who are pregnant, planning to become pregnant, or lactating.
* Requiring any change in doses of cardiovascular medication (including diuretics) in order to control worsening of HF symptoms.
* Known allergy to gadolinium.
* Currently receiving treatment with therapeutic doses of anticoagulants. Antiplatelet therapy used to prevent cardiovascular disease (primary prevention) or to treat chronic disease (secondary prevention) is permitted.
* Currently receiving treatment with sacubitril/valsartan or trimetazidine.
* Hyponatremia defined as plasma Na+ level <125 mEq/L (UK only).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerasimos Filippatos, MD, Study Chair — University of Athens, School of Medicine, Athens, Greece
Locations (15):
- Italy (8):
  - A.O. Papa Giovanni XXIII Cardiologia 1, Torre 5, Bergamo
  - A.O. Spedali Civili di Brescia Cardiologia, Brescia
  - Azienda Ospedaliera Brotzu Cardiologia, Cagliari
  - Centro Cardiologico Monzino U.O. Scompenso, Cardiologia Clinica e Cardiologia Riabilitativa, Milan
  - Ospedale Niguarda Ca' Granda SC Cardiologia 2, Milan
  - Cardiologia clinica, Unità dello Scompenso e Terapia intensive Reparto Carlo Magno, Faggi Policlinico di Monza, Monza
  - Dip. Cardiotoracovascolare: Cardiologia Fondazione IRCCS Policlinico San Matteo Pad. Nuovo Ospedale "DEA" Degenza: PIANO +3 Ambulatori: P.T. e P+3, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanità Pubblica, Pisa
- Netherlands (5):
  - Deventer Hospital, Department of Cardiology, Deventer
  - University Medical Centre Groningen, Groningen
  - Anthonius Ziekenhuis, Cardiology Department, Sneek
  - Elisabeth Twee Steden Hospital (ETZ), Department of Cardiology, Tilburg
  - Gelre Ziekenhuis Zutphen, Department of Cardiology, Zutphen
- United Kingdom (2):
  - Ninewells Hospital and Medical School, Dundee
  - William Harvey Heart Centre CRC, (Barts Health NHS Trust), London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Started | 23 | 24 | 24
Completed | 22 | 24 | 24
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 22 subjects in the 4 mg group, 1 subject (1.4%) discontinued from the study due to an AE. One of the subjects randomized to 4mg elamipretide arm was treated with 40mg elamipretide.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo | Total
Number analyzed (Participants) | 22 | 25 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.76) | 62.6 (9.63) | 66.8 (9.07) | 64.8 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 9 | 17
  Male | 19 | 20 | 15 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 24 | 24 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 25 | 24 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Left ventricular end systolic volume [Mean (Standard Deviation); unit: mL] — Left ventricular end systolic volume (ml) as measured by MRI
  mL | 87.0 (38.45) | 79.6 (21.54) | 77.7 (38.58) | 81.3 (33.28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End Systolic Volume (ml)
Description: Change in left ventricular end systolic volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom left ventricular end systolic volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Groups:
- 4 mg Elamipretide: 4 mg elamipretide: subcutaneous injection administered once daily for 28 consecutive days
- 40 mg Elamipretide: 40 mg elamipretide: subcutaneous injection administered once daily for 28 consecutive days
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
mL | -4.4 (6.50) | -1.2 (9.04) | -3.8 (5.85)

2. Secondary Outcome: Change in Left Ventricular Ejection Fraction (% of Blood Volume)
Description: Change in Left Ventricular Ejection Fraction as measured by percentage of blood volume from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for Left Ventricular Ejection Fraction was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
percentage of blood volume | 2.2 (2.43) | 1.5 (2.82) | 2.3 (3.69)

3. Secondary Outcome: Change in Left Ventricular End Diastolic Volume (ml) as Measured by MRI
Description: Change from baseline in Left Ventricular End Diastolic Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular End Diastolic Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
mL | -2.8 (9.50) | 0.5 (11.96) | -2.2 (9.77)

4. Secondary Outcome: Change in Left Ventricular Stroke Volume (ml)
Description: Change in Left Ventricular Stroke Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular Stroke Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
mL | 3.1 (9.23) | 3.7 (9.36) | 3.0 (13.14)

5. Secondary Outcome: Change in Left Ventricular Cardiac Output (L/Min)
Description: Change in Left Ventricular Cardiac Output as measured by L/min from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular Cardiac Output was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
L/min | 0.21 (1.264) | -0.01 (1.004) | 0.27 (0.860)

6. Secondary Outcome: Change in Left Ventricular Myocardial Mass (g)
Description: Change in Left Ventricular Myocardial Mass as measured by grams from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular Myocardial Mass was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
grams | 0.0 (2.82) | -0.4 (2.78) | -0.0 (2.26)

7. Secondary Outcome: Change in Right Ventricular End Systolic Volume (mL)
Description: Change in Right Ventricular End Systolic Volume as measured by mL from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Right Ventricular End Systolic Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
mL | -0.9 (4.21) | -0.8 (4.94) | -0.6 (3.72)

8. Secondary Outcome: Change in Right Ventricular End Diastolic Volume (mL)
Description: Change in Right Ventricular End Diastolic Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Right Ventricular End Diastolic Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
mL | 0.5 (9.70) | -1.2 (10.72) | -0.0 (7.61)

9. Secondary Outcome: Change in Right Ventricular Ejection Fraction (% Blood Volume)
Description: Change in Right Ventricular Ejection Fraction as measured by percentage of blood volume from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by MRI.
Time Frame: Baseline to Week 4
Population: All participants for whom Right Ventricular Ejection Fraction was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 22 | 24 | 23
percentage of blood volume | 1.4 (3.05) | 0.4 (2.10) | 1.2 (3.33)

10. Secondary Outcome: Change in Early and Late Mitral Inflow Velocity Ratio
Description: Change in Early and Late Mitral Inflow Velocity Ratio from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Early and Late Mitral Inflow Velocity Ratio was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 20 | 23 | 22
ratio | -0.04 (0.185) | -0.03 (0.329) | -0.07 (0.528)

11. Secondary Outcome: Change in Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity Ratio (E/e')
Description: Change in Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity Ratio as measured by E/e' from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity Ratio was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 21 | 23 | 22
ratio | -0.94 (3.244) | 0.47 (4.359) | -0.20 (4.287)

12. Secondary Outcome: Change in Left Atrial Volume (mL)
Description: Change in Left Atrial Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Atrial Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 20 | 20 | 22
mL | -3.4 (6.85) | -0.2 (4.41) | 1.6 (4.02)

13. Secondary Outcome: Change in Left Ventricular Global Longitudinal Strain Assessment (%)
Description: Change in Left Ventricular Global Longitudinal Strain Assessment as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular Global Longitudinal Strain Assessment was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: percentage of myocardial length change
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 4 | 3 | 9
percentage of myocardial length change | -1.76 (1.993) | -1.50 (2.721) | -1.46 (2.362)

14. Secondary Outcome: Change in Left Ventricular End Diastolic Volume (mL) as Measured by Echocardiography
Description: Change in Left Ventricular End Diastolic Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular End Diastolic Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 15 | 16 | 20
mL | -1.1 (16.29) | 1.6 (13.68) | 2.0 (15.29)

15. Secondary Outcome: Change in Left Ventricular End Systolic Volume (mL) as Measured by Echocardiography
Description: Change in Left Ventricular End Systolic Volume as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular End Systolic Volume was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 15 | 16 | 20
mL | -1.9 (11.59) | -0.5 (7.91) | 0.6 (10.31)

16. Secondary Outcome: Change in Biplane Ejection Fraction (mL)
Description: Change in Biplane Ejection Fraction as measured by ml from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Biplane Ejection Fraction was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 14 | 16 | 20
mL | 1.8 (2.94) | 2.0 (2.82) | 1.5 (4.22)

17. Secondary Outcome: Left Ventricular Mass Assessment (g)
Description: Change in Left Ventricular Mass Assessment as measured by grams from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Left Ventricular Mass was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 15 | 15 | 20
grams | 3.0 (18.26) | -4.2 (18.55) | -0.7 (21.99)

18. Secondary Outcome: Change in Tricuspid Regurgitation Severity Assessment (cm²)
Description: Change in Tricuspid Regurgitation Severity Assessment as measured by cm from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Tricuspid Regurgitation Severity Assessment was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 2 | 2 | 1
cm² | -1.03 (1.334) | 0.25 (1.336) | -0.30

19. Secondary Outcome: Change in Right Ventricular Fractional Area (%)
Description: Change Right Ventricular Fractional Area in as measured by percentage from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Right Ventricular Fractional Area was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: percentage of area
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 13 | 14 | 15
percentage of area | 0.1 (10.82) | 0.1 (8.79) | 0.9 (8.93)

20. Secondary Outcome: Change in Right Ventricular Systolic Pressure (mmHg)
Description: Change in Change in Right Ventricular Systolic Pressure as measured by mmHg from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Right Ventricular Systolic Pressure was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 8 | 9 | 8
mmHg | 5.7 (16.19) | -1.5 (6.63) | -7.0 (25.61)

21. Secondary Outcome: Change in Mitral Regurgitation Severity (cm²)
Description: Change in Mitral Regurgitation Severity as measured by cm² from baseline (last assessment prior to start of study) to Week 4 (end of treatment visit) as assessed by echocardiography.
Time Frame: Baseline to Week 4
Population: All participants for whom Mitral Regurgitation Severity was measured at baseline and Week 4
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
Number analyzed (Participants) | 5 | 5 | 6
cm² | 0.70 (2.668) | -0.71 (2.200) | -0.73 (1.834)

ADVERSE EVENTS:
Time Frame: 10 weeks (The AE reporting period began when the subject signed the ICF and continued through the clinical study's post treatment follow-up period, defined as 14 days after last administration of study medication.)
Arm/Group | 4 mg Elamipretide | 40 mg Elamipretide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/25 | 0/24
Other Adverse Events (participants affected / at risk) | 9/22 | 16/25 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg Elamipretide (N=22) | 40 mg Elamipretide (N=25) | Placebo (N=24)
Vestibular (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg Elamipretide (N=22) | 40 mg Elamipretide (N=25) | Placebo (N=24)
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Increased Blood bilirubin (Investigations) | 0 | 1 | 0
Eosinphil count increased (Investigations) | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 0
Injection site mass (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Insomia (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Albuminiuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02788747/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT02788747/SAP_001.pdf